CLINICAL TRIAL: NCT05845320
Title: Prevalence of Stress Urinary Incontinence in Obese Versus Non-obese Nulligravid Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS 188/2023
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese: BMI>30
  Interventions: Other: ICIQ-UI SF questionnaire
- Non-obesse: BMI<25
  Interventions: Other: ICIQ-UI SF questionnaire

INTERVENTIONS:
Other: ICIQ-UI SF questionnaire — validated arabic short form of ICIQ on urinary incontinence

SUMMARY:
Urinary incontinence (UI) is more common than any other chronic disease. Stress urinary incontinence (SUI), among the various forms of urinary incontinence, is the most prevalent (50%) type of this condition. Female urinary continence is maintained through an integrated function of pelvic floor muscles (PFMs), fascial structures, nerves, supporting ligaments, and the vagina. In women with SUI, the postural activity of the PFMs is delayed, and the balance ability is decreased. Many women, by learning the correct timing of a pelvic floor contraction during a cough, are able to eliminate consequent SUI. Timing is an important function of motor coordination and could be affected by proprioception.

We aim to assess stress urinary incontinence in obese and non-obese Nulligravid females.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between18 and 45 years.
* Non obese females with BMI <25kg/m2.
* Obese females with BMI ≥30kg/m2.
* Nulligravid females.

Exclusion Criteria:

* Multiparous Females
* Patients with active urinary tract infection.
* Patients with respiratory or neurological diseases.
* Patients with communication problems, cognitive disorders & mental disturbance.
* Current treatment with drugs (benzodiazepines, diuretics)
* Patients who underwent any previous abdominal or pelvic surgery.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: healthy nulligravid females
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Stress Urinary Incontinence in Obese Versus Non-obese Nulligravid Women | 6 months
  as detected by questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Maii Nawara, MD, Principal Investigator — Associate professor
Locations (1):
- Ain Shams University maternity hospital, Cairo, Cairo/القاهرة, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be available with principal investigator upon request